CLINICAL TRIAL: NCT05602727
Title: A Phase 2a/2b Randomized, Placebo-Controlled Clinical Study To Evaluate The Safety And Efficacy Of MK-1942 As Adjunctive Therapy In Participants With Mild To Moderate Alzheimer's Disease Dementia
Brief Title: Efficacy and Safety of MK-1942 as an Adjunct Therapy in Participants With Mild to Moderate Alzheimer's Disease Dementia (MK-1942-008)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Voluntarily terminated due to benefit/risk assessment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1942-008; MK-1942-008 (Other: MSD Protocol Number); jRCT2031220532 (Registry Identifier: jRCT); 2021-006336-94 (EudraCT Number)
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-1942 5 mg (Experimental): Participants will receive a single 5 mg MK-1942 capsule twice daily (BID), taken orally for 12 weeks. A mock titration will be done to maintain the study blind despite no changes in dose.
  Interventions: Drug: MK-1942
- MK-1942 15 mg (Experimental): Participants will receive a single 8 mg MK-1942 capsule twice daily (BID), taken orally for one week. Then the dose is titrated up to 15 mg MK-1942 capsule twice daily (BID), taken orally for up to 11 weeks.
  Interventions: Drug: MK-1942
- Placebo (Placebo Comparator): Participants will receive a placebo capsule twice daily (BID), taken orally for 12 weeks. A mock titration will be done to maintain the study blind despite no changes in dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-1942 — MK-1942 oral capsule
  Arms: MK-1942 15 mg; MK-1942 5 mg
Drug: Placebo — Placebo oral capsule
  Arms: Placebo

SUMMARY:
The main purpose of this study was to assess the safety and efficacy of MK-1942 as adjunctive therapy in participants with mild to moderate Alzheimer's Disease (AD) dementia.

ELIGIBILITY:
Inclusion Criteria:

* Has mild to moderate AD dementia based on the national institute of neurological and communicative diseases and stroke/Alzheimer's Disease and related disorders association (NINCDS-ADRDA) criteria.
* Has mini-mental state examination (MMSE) score between 12-22 (inclusive) at screening.
* Is using acetylcholinesterase inhibitors (AChEI) therapy for management of AD dementia at Screening and during the study. These medications must be at stable approved dose levels ≥3 months before the first dose of study intervention and the regimens must remain constant throughout the study to the extent that is clinically appropriate.
* Has a designated study partner who can fulfill the requirements of this study. The study partner will need to spend sufficient time with the participant to be familiar with their overall function and behavior and be able to provide adequate information about the participant needed for the study including, knowledge of functional and basic activities of daily life, work/educational history, cognitive performance, emotional/psychological state, and general health status.

Exclusion Criteria:

* Has a known history of stroke or cerebrovascular disease that is clinically important in the investigator's opinion.
* Has diagnosis of a clinically relevant central nervous system (CNS) disease other than AD dementia (with protocol-specified exceptions).
* Has a history of seizures or epilepsy within the 10 years preceding Screening.
* Has any other major CNS trauma, or infections that affect brain function.
* Has evidence of a clinically relevant or unstable psychiatric disorder, based on criteria from the diagnostic and statistical manual of mental disorders (fifth edition), including schizophrenia or other psychotic disorder, bipolar disorder, major depression, or delirium. Major depression in remission is not exclusionary.
* Has a severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or administration intervention.
* Has a history of malignancy occurring within the 5 years immediately before Screening, except for a participant who has been adequately treated for 1 or more of the following: basal cell or squamous cell skin cancer; in situ cervical cancer; localized prostate carcinoma; who has undergone potentially curative therapy with no evidence of recurrence for ≥3 years post-therapy, and who is deemed to be at low risk for recurrence.
* Has a risk factor for QTc prolongation.
* Has a history of alcoholism or drug dependency/abuse within the 5 years preceding screening.
* Has a known allergy or intolerance to the active or inert ingredients in MK-1942.
* Has received any anti-amyloid agents or antibodies, or any of the following medications: CNS-penetrant anticholinergics, neuroleptics, anticonvulsants, narcotics, glutamatergic agents, agents with possible psychotropic effects, and experimental acute respiratory syndrome coronavirus 2 (COVID-19) therapies.
* Has liver disease, including but not limited to chronic viral hepatitis, non viral hepatitis, cirrhosis, malignancies, autoimmune liver diseases.
* Has an abnormal thyroid-stimulating hormone (TSH) value if confirmed by abnormal T4 value.
* Resides in a nursing home or assisted care facility with need for direct continuous medical care and nursing supervision. Participant may reside in such facilities provided continuous direct medical care is not required and a qualified study partner is available for coparticipation and the participant is physically able to attend all required study visits.
* Had major surgical procedure or donated or lost >1 unit of blood (approximately 500 mL) within the 4 weeks before screening.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (74):
- United States (22):
  - Banner Alzheimer's Institute ( Site 0017), Phoenix, Arizona
  - Neurology Center of North Orange County ( Site 0039), Fullerton, California
  - California Neuroscience Research, LLC ( Site 0058), Sherman Oaks, California
  - JEM Research Institute ( Site 0013), Atlantis, Florida
  - Velocity Clinical Research, Hallandale Beach ( Site 0025), Hallandale, Florida
  - K2 Medical Research ( Site 0057), Maitland, Florida
  - Premier Clinical Research Institute ( Site 0038), Miami, Florida
  - Collier Neurologic Specialists ( Site 0045), Naples, Florida
  - Atlanta Center for Medical Research ( Site 0044), Atlanta, Georgia
  - iResearch Atlanta ( Site 0016), Decatur, Georgia
  - Alexian Brothers Medical Center ( Site 0011), Elk Grove Village, Illinois
  - Tandem Clinical Research ( Site 0055), Marrero, Louisiana
  - Global Medical Institutes LLC; Princeton Medical Institute ( Site 0053), Princeton, New Jersey
  - Advanced Memory Research Institute of New Jersey ( Site 0027), Toms River, New Jersey
  - Richmond Behavioral Associates ( Site 0008), Staten Island, New York
  - AMC Research, LLC ( Site 0004), Matthews, North Carolina
  - NeuroScience Research Center ( Site 0009), Canton, Ohio
  - Summit Headlands ( Site 0018), Portland, Oregon
  - Grayline Research Center ( Site 0003), Wichita Falls, Texas
  - The Memory Clinic ( Site 0054), Bennington, Vermont
  - Re:Cognition Health ( Site 0031), Fairfax, Virginia
  - Northwest Clinical Research Center ( Site 0056), Bellevue, Washington
- Argentina (6):
  - Clinica Privada Banfield ( Site 0205), Banfield, Buenos Aires
  - Hospital Italiano de Buenos Aires-Geriatrics ( Site 0210), Buenos Aires, Buenos Aires F.D.
  - Instituto Kremer ( Site 0202), Córdoba, Córdoba Province
  - IDIM - Instituto de Diagnóstico e Investigaciones Metabólicas ( Site 0204), Buenos Aires
  - Instituto Geriatrico Nuestra Señora de Las Nieves ( Site 0208), Buenos Aires
  - Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (FLENI) ( Site 0201), Buenos Aires
- Australia (3):
  - KARA Institute for Neurological Diseases ( Site 1902), Sydney, New South Wales
  - Austin Health-Medical & Cognitive Research Unit ( Site 1901), Ivanhoe, Victoria
  - HammondCare ( Site 1903), Malvern, Victoria
- Canada (6):
  - OCT Research ULC ( Site 0113), Kelowna, British Columbia
  - Centricity Research - Halifax ( Site 0111), Halifax, Nova Scotia
  - Ottawa Memory Clinic ( Site 0105), Ottawa, Ontario
  - Sunnybrook Health Sciences Centre ( Site 0106), Toronto, Ontario
  - Toronto Western Hospital-Memory clinic ( Site 0102), Toronto, Ontario
  - Clinique de la Mémoire de l'Outaouais ( Site 0114), Gatineau, Quebec
- Colombia (4):
  - Instituto Neurológico de Colombia ( Site 0415), Medellín, Antioquia
  - Grupo Neurociencias de Antioquia ( Site 0417), Medellín, Antioquia
  - Centro de Investigaciones del Sistema Nervioso - Grupo Cisne ( Site 0414), Bogotá, Bogota D.C.
  - Fundacion Valle del Lili- CIC ( Site 0418), Cali, Valle del Cauca Department
- Italy (5):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore (, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico-UOSD Malattie Neurodegenerative ( Site 1204, Milan, Lombardy
  - Ospedale San Raffaele ( Site 1202), Milan, Lombardy
  - Ospedale San Gerardo-ASST Monza-Dipartimento di Neuroscienze ( Site 1201), Monza, Lombardy
  - Centro S Giovanni Di Dio Fatebenefratelli ( Site 1205), Brescia
- Japan (8):
  - Kakigi Cognition and Emotion Clinic of Hope ( Site 2307), Kobe, Hyōgo
  - Kagawa University Hospital ( Site 2308), Kita-gun, Kagawa-ken
  - Kishiro Mental Clinic ( Site 2310), Kawasaki, Kanagawa
  - Kawasaki Saiwai Clinic ( Site 2302), Saiwaiku,Kawasaki, Kanagawa
  - Nagomi Clinic ( Site 2305), Toyonaka, Osaka
  - Tokyo Metropolitan Geriatric Hospital ( Site 2301), tabashi City, Tokyo
  - Ishikawa Clinic ( Site 2306), Kyoto
  - Himuro Neurology Clinic ( Site 2304), Osaka
- CGM Research Trust ( Site 2001), Christchurch, Canterbury, New Zealand
- South Korea (4):
  - Inha University Hospital ( Site 2104), Incheon
  - Asan Medical Center-Department of Neurology ( Site 2101), Seoul
  - Samsung Medical Center ( Site 2102), Seoul
  - Ewha Womans University Seoul Hospital ( Site 2103), Seoul
- Spain (9):
  - Hospital Universitari Mutua Terrassa-Neurology ( Site 1607), Terrassa, Barcelona
  - Centro de Atención Especializada Oroitu ( Site 1610), Getxo, Basque Country
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 1609), Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau ( Site 1603), Barcelona, Catalonia
  - Clinica Universidad de Navarra-Neurology ( Site 1602), Pamplona, Navarre
  - Hospital Universitario Doctor Peset-Neurología ( Site 1601), Valencia, Valenciana, Comunitat
  - Fundació ACE ( Site 1604), Barcelona
  - Hospital Clinico San Carlos ( Site 1608), Madrid
  - Hospital Viamed Montecanal-Neurociencia ( Site 1606), Zaragoza
- United Kingdom (6):
  - Brain Health Scotland Life Sciences ( Site 1810), Edinburgh, Edinburgh, City of
  - Queen Elizabeth University Hospital-Glasgow Clinical Research Facility ( Site 1808), Glasgow, Glasgow City
  - Re:Cognition Health - London ( Site 1804), London, London, City of
  - Kingshill Research Centre ( Site 1807), Swindon, Wiltshire
  - Re:Cognition Health - Birmingham ( Site 1801), Birmingham
  - Re:Cognition Health - Plymouth ( Site 1803), Plymouth

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26357&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled at study sites located in USA, UK, Spain, Japan, Republic of Korea, Canada, Argentina, and Australia.
Groups:
- MK-1942 5 mg: Participants received MK-1942 5 mg twice daily (BID) for 12 weeks without dose titration.
- MK-1942 15 mg: Participants received MK-1942 8 mg BID for 1 week, followed by MK-1942 15 mg BID for the next 11 weeks.
- Placebo: Participants received an inert placebo matched to MK-1942 BID for 12 weeks.
Period: Overall Study
Arm/Group | MK-1942 5 mg | MK-1942 15 mg | Placebo
Started | 35 | 31 | 33
Completed | 13 | 8 | 12
Not Completed | 22 | 23 | 21
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Randomized by mistake without study medication | 1 | 0 | 0
Not completed — Study termination by Sponsor | 18 | 15 | 19
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Various reasons | 1 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1942 5 mg | MK-1942 15 mg | Placebo | Total
Number analyzed (Participants) | 35 | 31 | 33 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.1 (7.5) | 74.7 (8.0) | 72.3 (8.2) | 73.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 23 | 69
  Male | 10 | 10 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 2 | 10
  Not Hispanic or Latino | 33 | 25 | 31 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 29 | 28 | 26 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Alzheimer's Disease Assessment Scale-11-item Cognitive Subscale (ADAS-Cog11) Score at Week 12
Description: The change from baseline in ADAS-Cog11 score is presented. ADAS-Cog11 is a structured scale that evaluates memory, orientation, attention, reasoning, language, and constructional praxis. ADAS-Cog11 measures cognition by assessing 11 metrics impaired in AD: word recall; commands; constructional praxis; naming objects and fingers; ideational praxis; orientation; word recognition; remembering test instructions; spoken language ability; word-finding difficulty; and comprehension of spoken language. The total possible score ranges from 0 to 70, with higher scores indicating greater cognitive impairment. Negative values indicate improvement relative to baseline, and vice versa.
Time Frame: Baseline and Week 12
Population: Randomized participants who received ≥1 dose of study treatment, and who have baseline and a post-baseline assessment available, are included. A mixed-model repeated measures analyses was used in which partial data from participants not completing the study was utilized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- MK-1942 5 mg: Participants received MK-1942 5 mg BID for 12 weeks without dose titration.
Arm/Group | MK-1942 5 mg | MK-1942 15 mg | Placebo
Number analyzed (Participants) | 20 | 21 | 25
Units on a scale | 2.9 [0.7 to 5.1] | -0.6 [-3.0 to 1.8] | 0.8 [-1.4 to 3.0]
Statistical Analysis 1: Comparison: MK-1942 5 mg vs Placebo; Test type: Superiority — Difference in LS Means (MK-1942 - Placebo); p = 0.186, Longitudinal ANCOVA; LS Mean Difference = 2.1, 97.5% CI 2-sided [-1.6 to 5.8]
Statistical Analysis 2: Comparison: MK-1942 15 mg vs Placebo; Test type: Superiority — Difference in LS Means (MK-1942 - Placebo); p = 0.400, Longitudinal ANCOVA; LS Mean Difference = -1.4, 97.5% CI 2-sided [-5.2 to 2.4]

2. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to ~ 14 Weeks
Population: All randomized participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1942 5 mg | MK-1942 15 mg | Placebo
Number analyzed (Participants) | 34 | 31 | 33
Participants | 17 | 21 | 18

3. Primary Outcome: Number of Participants Discontinuing Study Medication Due to an Adverse Event
Description: as for outcome 2
Time Frame: Up to ~ 12 Weeks
Population: All participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1942 5 mg | MK-1942 15 mg | Placebo
Number analyzed (Participants) | 34 | 31 | 33
Participants | 4 | 6 | 3

4. Secondary Outcome: Alzheimer's Disease Cooperative Study Clinical Global Impression of Change (ADCS-CGIC) Overall Score at Week 12
Description: The overall score in ADCS-CGIC is presented. ADCS-CGIC is a global scale assessing cognition and function based on structured interviews of both the participant and study partner. ADCS-CGIC focuses on clinicians' observations of change in the patient's cognitive, functional, and behavioral performance since the beginning of the study. Improvement in the ADCS-CGIC overall score, with a score of 1, 2, or 3 indicates improvement. The ADCS-CGIC is a clinician-rated measure of global severity at baseline scored from 1 (normal, not at all ill) to 7 (among the most extremely ill patients); and global change at follow-up scored from 1 (marked improvement) to 7 (marked worsening), where 4 indicates no change.
Time Frame: Week 12
Population: Randomized participants who received ≥1 dose of study treatment, and who have the relevant assessment available, are included.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MK-1942 5 mg | MK-1942 15 mg | Placebo
Number analyzed (Participants) | 14 | 11 | 13
Units on a scale | 5.4 (0.7) | 5.8 (0.9) | 5.3 (0.8)

5. Secondary Outcome: Mean Change From Baseline in The Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) Total Score at Week 12
Description: The change from baseline in ADCS-ADL score is presented. The ADCS-ADL is an informant-based measure of the participant's functional ability in activities of daily living. The ADCS-ADL assesses the competence of participants with AD dementia in basic and instrumental ADLs. The ADCS-ADL is a 23-item scale that includes 6 basic ADL items and 17 instrumental ADL items that provide a total score ranging from 0 to 78, with a lower score indicating greater severity.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | MK-1942 5 mg | MK-1942 15 mg | Placebo
Number analyzed (Participants) | 20 | 21 | 25
Units on a scale | -1.7 [-4.8 to 1.4] | -3.0 [-6.4 to 0.4] | 1.2 [-2.0 to 4.4]
Statistical Analysis 1: Comparison: MK-1942 5 mg vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.196, Longitudinal ANCOVA; LS Mean Difference = -2.9, 97.5% CI 2-sided [-8.0 to 2.2]
Statistical Analysis 2: Comparison: MK-1942 15 mg vs Placebo; Test type: Superiority — Difference in LS Means; p = 0.081, Longitudinal ANCOVA; LS Mean Difference = -4.2, 97.5% CI 2-sided [-9.6 to 1.3]

ADVERSE EVENTS:
Time Frame: Up to ~14 weeks
Description: All participants who received ≥1 dose of study treatment are included.
Arm/Group | MK-1942 5 mg | MK-1942 15 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/34 | 2/31 | 2/33
Other Adverse Events (participants affected / at risk) | 16/34 | 16/31 | 12/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-1942 5 mg (N=34) | MK-1942 15 mg (N=31) | Placebo (N=33)
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-1942 5 mg (N=34) | MK-1942 15 mg (N=31) | Placebo (N=33)
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1
Fatigue (General disorders) | 1 | 2 | 1
Feeling abnormal (General disorders) | 2 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 4
Alanine aminotransferase increased (Investigations) | 10 | 5 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 4 | 5 | 4
Headache (Nervous system disorders) | 3 | 1 | 1
Hypertension (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT05602727/Prot_SAP_000.pdf